CLINICAL TRIAL: NCT02997202
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase III Trial of the FLT3 Inhibitor Gilteritinib Administered as Maintenance Therapy Following Allogeneic Transplant for Patients With FLT3/ITD AML
Brief Title: A Trial of the FMS-like Tyrosine Kinase 3 (FLT3) Inhibitor Gilteritinib Administered as Maintenance Therapy Following Allogeneic Transplant for Patients With FLT3/Internal Tandem Duplication (ITD) Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2215-CL-0304; 2016-001061-83 (EudraCT Number); BMT CTN 1506 (Other: Blood and Marrow Transplant Clinical Trials Network)
Expanded Access: NCT03070093 (Approved for marketing)
Record Dates: First submitted 2016-12-01; First posted 2016-12-19 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Gilteritinib; ASP2215; Safety and Efficacy; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gilteritinib (Experimental): Participants received gilteritinib 120 milligrams (mg) (three tablets of 40 mg) orally, once daily (QD) for up to 2 years or until a protocol-defined discontinuation criterion was met.
  Interventions: Drug: gilteritinib
- Placebo (Placebo Comparator): Participants received gilteritinib matching placebo orally, QD for up to 2 years or until a protocol-defined discontinuation criterion was met.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: gilteritinib — oral
  Arms: Gilteritinib
Drug: Placebo — oral
  Arms: Placebo

SUMMARY:
The purpose of this study was to compare relapse-free survival between participants with FLT3/ITD AML in first morphologic complete remission (CR1) who underwent hematopoietic stem cell transplant (HCT) and were randomized to receive gilteritinib or placebo beginning after the time of engraftment for a two year period.

DETAILED DESCRIPTION:
Participants with FLT3/ITD AML in first morphologic complete remission (CR1) undergone allogeneic hematopoietic stem cell transplant (HCT) were randomized to receive gilteritinib or placebo 30 to 90 days after HCT for a two year period. Participants wiere stratified according to: 1) conditioning regimen intensity (myeloablative vs. reduced intensity/non-myeloablative), 2) time from first day of hematopoietic cell infusion to randomization (30-60 days vs. 61-90 days) and 3) presence vs absence of or unknown minimal residual disease (MRD) from the most recent pre-registration bone marrow (BM) aspirate.

ELIGIBILITY:
Registration Inclusion Criteria

* Participant is considered a suitable candidate for HCT and has an acceptable source of allogeneic donor stem cells, as defined per institutional practice (allogeneic HCT for any donor source [matched sibling, unrelated donor (URD), mismatched URD, related haploidentical, or umbilical cord blood] and any graft source [umbilical cord, BM, peripheral blood (PB)], and any conditioning [myeloablative conditioning (MAC), reduced intensity conditioning (RIC), or non-myeloablative conditioning (NMA)] will be permitted).
* Participant is considered a legal adult by local regulation at the time of signing informed consent form (ICF).
* Participant consents to allow access to diagnostic BM aspirate or PB sample and/or the DNA derived from that sample, if available, that may be used to validate a companion diagnostic that is being developed in parallel with gilteritinib.
* Participant has confirmed, morphologically documented AML in CR1. For the purposes of registration, CR1 will be defined as < 5% blasts in the BM with no morphologic characteristics of acute leukemia (e.g., Auer Rods) in the BM with no evidence of extramedullary disease such as central nervous system involvement or granulocytic sarcoma.

  * Participant has not received more than 2 cycles of induction chemotherapy to achieve CR1. The induction cycles can be the same regimen or different regimens. The regimen(s) may contain conventional agents, investigational agents, or a combination of both.
  * Participants with CR with incomplete count recovery (CRp or CRi) are allowed. Incomplete platelet recovery (CRp) is defined as CR with platelet count < 100 x 109/L. Incomplete blood count recovery (CRi) is defined as CR with residual neutropenia < 1 x 109/L with or without complete platelet recovery. Red blood cell count (RBC) and platelet transfusion independence is not required.
  * The maximum time allowed from establishment of CR1 to registration is 12 months.
* Participant has presence of the FLT3/ITD activating mutation in the BM or PB as determined by the local institution at diagnosis.
* Participant must meet the following criteria as indicated on the clinical laboratory tests:

  * Serum creatinine within normal range, or if serum creatinine outside normal range, then glomerular filtration rate (GFR) > 40 mL/min/1.73m2 as calculated with the Cockcroft-Gault equation with adjustment if total body weight is ≥ 125% of ideal body weight.
  * Total bilirubin (TBL) ≤ 2.5 mg/dL, except for participants with Gilbert's syndrome.
  * Serum AST and/or alanine aminotransferase (ALT) < 3 x institutional upper limit of normal (ULN).
* Participant has left ventricular ejection fraction at rest ≥ 40%.
* Participant has diffusing capacity of the lung for carbon monoxide (DLCO) (corrected for hemoglobin) ≥ 50% predicted and/or forced expiratory volume in 1 second (FEV1) ≥ 50% predicted.
* Female participants must either:

  * Be of non-childbearing potential:
  * postmenopausal (defined as at least 1 year without menses) prior to screening or
  * documented as surgically sterilized (at least 1 month prior to the screening visit)
* Or, if of childbearing potential,

  * Agree not to try to become pregnant during the study for 6 months after the final study drug administration
  * And have a negative serum pregnancy test at screening
  * And, if heterosexually active, agree to consistently use highly effective contraception per locally accepted standards in addition to a barrier method starting at screening and throughout the study period and for 6 months after the final study drug administration.
  * For United Kingdom sites:
  * Highly effective forms of birth control include:
  * Consistent and correct usage of established hormonal contraceptives that inhibit ovulation
  * Established intrauterine device (IUD) or intrauterine system (IUS)
* Female participants must agree not to breastfeed or donate ova throughout the study drug treatment period and for 6 months after the final study drug administration.
* Male participants (even if surgically sterilized), and partners who are women of childbearing potential must be using highly effective contraception in addition to a barrier method throughout the study drug treatment period and for 127 days after the final study drug administration.

  * For United Kingdom sites:
  * Highly effective forms of birth control include:
  * Consistent and correct usage of established hormonal contraceptives that inhibit ovulation
  * Established IUD or IUS
  * Vasectomy (A vasectomy is a highly effective contraception method provided the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.)
  * Male is sterile due to a bilateral orchiectomy
* Male participants must not donate sperm throughout the study drug treatment period and for 127 days after the final study drug administration.
* Participant is able to take an oral medication.
* Participant agrees not to participate in another interventional study while on treatment.

Randomization Inclusion Criteria

* Participant is ≥ 30 days and ≤ 90 days from hematopoietic cell infusion.
* Participant has achieved engraftment. Engraftment is defined as ANC ≥ 500 cells/μL and platelets ≥ 20000/μL on 3 consecutive measurements (each occurring at least 1 day apart). The participant must not have had a platelet transfusion within 7 days prior to the first measurement.
* Participant has confirmed ongoing morphologically documented AML in CR1. For the purposes of randomization, CR1 will be defined as < 5% blasts with no morphologic characteristics of acute leukemia (e.g., Auer Rods) in the BM with no evidence of extramedullary disease such as central nervous system involvement or granulocytic sarcoma.
* Participant meets the following criteria as indicated on the clinical laboratory tests:

  * Serum creatinine within normal range, or if serum creatinine outside normal range, then GFR > 40 mL/min/1.73m2 as calculated with the Cockcroft-Gault equation with adjustment if total body weight is ≥ 125% of ideal body weight.
  * TBL < 2.5 mg/dL, except for participants with Gilbert's syndrome.
  * Serum AST and/or ALT < 3 x institutional ULN.
  * Serum potassium and magnesium ≥ the institutional lower limit of normal (LLN).
* If the participant has developed overall grades II-IV acute GVHD, the following criteria must be met to be randomized:

  * No requirement of > 0.5 mg/kg of prednisone (or equivalent) daily dose within 1 week of randomization
  * No escalation of systemic immunosuppression in terms of increase of corticosteroids or addition of new agent / modality within 2 weeks of randomization. (Note that increasing calcineurin inhibitors or sirolimus to achieve therapeutic trough levels is allowed.) Topical skin and topical gastrointestinal steroids are allowed.
* Participant is able to take oral medication.

Registration Exclusion Criteria

* Participant has had a prior allogeneic transplant.
* Participant has Karnofsky performance status score < 70% .
* Participant requires treatment with concomitant drugs that are strong inducers of CYP3A within 14 days of start of study drug.
* Participant requires treatment with concomitant drugs that target serotonin 5-hydroxytryptamine receptor 1 (5HT1R) or 5-hydroxytryptamine receptor 2B (5HT2BR) or sigma nonspecific receptor with the exception of drugs that are considered absolutely essential for the care of the participant.
* Participant has a Fridericia-corrected QT interval (QTcF) > 450 msec (average of triplicate determinations) per central read.
* Participant has long QT Syndrome at screening.
* Participant has a known infection with human immunodeficiency virus (HIV).
* Participant has active hepatitis B infection as determined by NAAT or surface antigen assay. Participants who have acquired immunity from past exposure (HBcAb positive / HBsAb positive / HBsAg negative) are eligible.
* Participant has active hepatitis C infection as determined by NAAT. NAAT must be performed if the participant has positive serology for hepatitis C. Participants who have had past exposure and have no detectable virus either through spontaneous clearance or treatment are eligible.
* Participant has an uncontrolled infection. If a bacterial or viral infection is present, the participant must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to registration. If a fungal infection is present, the participant must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to registration.

  * Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection.
  * Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
* Participant has had a myocardial infarction within 6 months prior to registration or New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia.
* Participant has a serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Participant is breast feeding or pregnant.
* Participant has prior malignancies, except lobular breast carcinoma in situ, fully resected basal cell or squamous cell carcinoma of skin or treated cervical carcinoma in situ.

Cancer treated with curative intent ≥ 5 years previously will be allowed. Cancer treated with curative intent < 5 years previously will not be allowed.

Randomization Exclusion Criteria

* Participant requires treatment with concomitant drugs that are strong inducers of CYP3A within 14 days of starting study drug.
* Participant requires treatment with concomitant drugs that target serotonin 5HT1R or 5HT2BR or sigma nonspecific receptor with the exception of drugs that are considered by the investigator to be absolutely essential for the care of the participant and for which no acceptable alternative exists.
* Participant has a QTcF interval > 450 msec (average of triplicate determinations) by central read.
* Participant has a need for supplemental oxygen with the exception of using previously existing non-invasive continuous positive airway pressure (CPAP) at night.
* Participant has used investigational agents within 4 weeks of randomization.
* Participant has used experimental therapy for acute GVHD within 4 weeks of randomization. If unsure of the definition of "experimental", discussion with one of the protocol chairs is recommended.
* Participant has an uncontrolled infection. If a bacterial or viral infection is present, the participant must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to randomization. If a fungal infection is present, the participant must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to randomization.

  * Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection.
  * Persisting fever without other signs or symptoms will not be interpreted as progressing infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2023-01-07 (Actual); Study Completion 2023-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (118):
- United States (46):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic, Phoenix, Arizona
  - Virginia G Piper Cancer Center, Scottsdale, Arizona
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northside, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana Blood and Marrow Transplant, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland Medical Systems, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - University of Minnesota School of Medicine, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University Hospitals of Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, The, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Intermountain BMT, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Site AU61001, Liverpool
  - Site AU61002, Melbourne
  - Site AU61004, Westmead
- Belgium (2):
  - Site BE32003, Brussels
  - Site BE32004, Ghent
- Canada (2):
  - Site CA15004, Hamilton
  - Site CA15003, Montreal
- Denmark (2):
  - Site DK45002, Aarhus
  - Site DK45001, Copenhagen
- France (5):
  - Site FR33007, Lille
  - Site FR33004, Lyon
  - Site FR33005, Paris
  - Site FR33008, Pessac
  - Site FR33010, Vandœuvre-lès-Nancy
- Germany (6):
  - Site DE49006, Cologne
  - Site DE49002, Düsseldorf
  - Site DE49003, Halle
  - Site DE49005, Hamburg
  - Site DE49007, Mainz
  - Site DE49004, Münster
- Greece (3):
  - Site GR30004, Athens
  - Site GR30003, Rio
  - Site GR30001, Thessaloniki
- Italy (8):
  - Site IT39005, Bergamo
  - Site IT39006, Bologna
  - Site IT39009, Genova
  - Site IT39002, Milan
  - Site IT39007, Milan
  - Site IT39011, Pescara
  - Site IT39003, Roma
  - Site IT39004, Udine
- Japan (19):
  - Site JP81014, Anjo, Aichi-ken
  - Site JP81011, Nagoya, Aichi-ken
  - Site JP81018, Sapporo, Hokkaido
  - Site JP81021, Kobe, Hyōgo
  - Site JP81012, Nishinomiya, Hyōgo
  - Site JP81002, Isehara, Kanagawa
  - Site JP81007, Yokohama, Kanagawa
  - Site JP81010, Sendai, Miyagi
  - Site JP81006, Suita, Osaka
  - Site JP81008, Shimotsuke, Tochigi
  - Site JP81013, Bunkyo-ku, Tokyo
  - Site JP81004, Chuo-ku, Tokyo
  - Site JP81016, Minato-ku, Tokyo
  - Site JP81020, Shinjuku-ku, Tokyo
  - Site JP81001, Fukuoka
  - Site JP81003, Fukuoka
  - Site JP81015, Kyoto
  - Site JP81017, Okayama
  - Site JP81005, Osaka
- New Zealand (2):
  - Site NZ64002, Christchurch
  - Site NZ64001, Grafton
- Site PL48004, Warsaw, Poland
- South Korea (5):
  - Site KR82001, Seoul
  - Site KR82002, Seoul
  - Site KR82003, Seoul
  - Site KR82004, Seoul
  - Site KR82005, Seoul
- Spain (5):
  - Site ES34004, Barcelona
  - Site ES34005, Barcelona
  - Site ES34006, Salamanca
  - Site ES34007, Santander
  - Site ES34002, Valencia
- Taiwan (3):
  - Site TW88603, Taichung
  - Site TW88602, Taipei
  - Site TW88605, Taoyuan District
- United Kingdom (6):
  - Site GB44010, Birmingham
  - Site GB44003, Bristol
  - Site GB44009, Glasgow
  - Site GB44004, London
  - Site GB44002, Manchester
  - Site GB44001, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Levis MJ, Hamadani M, Logan BR, Jones RJ, Singh AK, Litzow MR, Wingard JR, Papadopoulos EB, Perl AE, Soiffer RJ, Ustun C, Oshima MU, Uy GL, Waller EK, Vasu S, Solh M, Mishra A, Muffly LS, Kim HJ, Stelljes M, Najima Y, Onozawa M, Thomson K, Chen C, Hasabou N, Rosales M, Hill JE, Gill SC, Nuthethi R, King D, Mendizabal A, Devine SM, Horowitz MM, Chen YB. Impact of transplant conditioning, NPM1 mutations, and measurable residual disease in FLT3-ITD acute myeloid leukemia. Blood Adv. 2025 Oct 28;9(20):5123-5133. doi: 10.1182/bloodadvances.2025016306. PMID 40590852
- [Derived] Levis MJ, Hamadani M, Logan BR, Jones RJ, Singh AK, Litzow MR, Wingard JR, Papadopoulos EB, Perl AE, Soiffer RJ, Ustun C, Oshima MU, Uy GL, Waller EK, Vasu S, Solh M, Mishra A, Muffly LS, Kim HJ, Stelljes M, Najima Y, Onozawa M, Thomson K, Nagler A, Wei AH, Marcucci G, Chen C, Hasabou N, Rosales M, Hill J, Gill SC, Nuthethi R, King D, Mendizabal A, Devine SM, Horowitz MM, Chen YB. Measurable residual disease and posttransplantation gilteritinib maintenance for patients with FLT3-ITD-mutated AML. Blood. 2025 May 8;145(19):2138-2148. doi: 10.1182/blood.2024025154. PMID 39775763
- [Derived] Hamilton BK, Pandya BJ, Ivanescu C, Elsouda D, Hamadani M, Chen YB, Levis MJ, Ueda Oshima M, Litzow MR, Soiffer RJ, Ustun C, Perl AE, Singh AK, Geller N, Hasabou N, Rosales M, Cella D, Corredoira L, Pestana C, Horowitz MM, Logan B. Health-related quality of life with gilteritinib vs placebo posttransplant for FLT3-ITD+ acute myeloid leukemia. Blood Adv. 2024 Oct 8;8(19):5091-5099. doi: 10.1182/bloodadvances.2024013746. PMID 39167766
- [Derived] Pandya BJ, Burns LJ, Wang T, Xie B, Touya M, Spalding J, Block A, Kuperman G, Young C. Clinical Outcomes and Treatment Patterns in Adults With FLT3-ITDmut+ Acute Myeloid Leukemia Undergoing Allogeneic Hemopoietic Cell Transplantation in the United States and Canada. Transplant Cell Ther. 2024 Jul;30(7):683.e1-683.e13. doi: 10.1016/j.jtct.2024.04.016. Epub 2024 Apr 23. PMID 38663769
- [Derived] Levis MJ, Hamadani M, Logan B, Jones RJ, Singh AK, Litzow M, Wingard JR, Papadopoulos EB, Perl AE, Soiffer RJ, Ustun C, Ueda Oshima M, Uy GL, Waller EK, Vasu S, Solh M, Mishra A, Muffly L, Kim HJ, Mikesch JH, Najima Y, Onozawa M, Thomson K, Nagler A, Wei AH, Marcucci G, Geller NL, Hasabou N, Delgado D, Rosales M, Hill J, Gill SC, Nuthethi R, King D, Wittsack H, Mendizabal A, Devine SM, Horowitz MM, Chen YB; BMT-CTN 1506/MORPHO Study Investigators. Gilteritinib as Post-Transplant Maintenance for AML With Internal Tandem Duplication Mutation of FLT3. J Clin Oncol. 2024 May 20;42(15):1766-1775. doi: 10.1200/JCO.23.02474. Epub 2024 Mar 12. PMID 38471061
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14519&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with FMS-like tyrosine kinase 3/Internal tandem duplication (FLT3/ITD) acute myeloid leukemia (AML) in first morphological complete remission (CR1) including complete remission with incomplete platelet recovery (CRp) & complete remission with incomplete hematologic recovery (CRi) undergoing allogeneic hematopoietic cell transplant (HCT) were enrolled in the study.
Pre-assignment Details: Randomization was stratified by: Conditioning regimen intensity myeloablative vs reduced intensity/non-myeloablative (RIC/NMA); Time from first day of hematopoietic cell infusion to randomization (30 to 60 vs 61 to 90 days); Presence vs absence of/unknown, Minimal Residual Disease-4 (MRD-4) from the most recent pre-registration Bone marrow (BM).
Period: Overall Study
Arm/Group | Gilteritinib | Placebo
Started | 178 (1 participant randomized to gilteritinib did not take any gilteritinib or placebo) | 178 (1 participant randomized to placebo took gilteritinib)
Safety Analysis Population | 178 | 177
Intent to Treat (ITT) Population | 178 | 178
Completed | 122 | 116
Not Completed | 56 | 62
Not completed — Miscellaneous | 2 | 2
Not completed — Withdrawal by Subject | 8 | 12
Not completed — Lost to Follow-up | 5 | 3
Not completed — Death | 41 | 45

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat (ITT) population: All randomized participants were included in this population
Groups:
- Gilteritinib: Participants received gilteritinib 120 mg (three tablets of 40 mg) orally, QD for up to 2 years or until a protocol-defined discontinuation criterion was met.
- Total: Total of all reporting groups
Arm/Group | Gilteritinib | Placebo | Total
Number analyzed (Participants) | 178 | 178 | 356
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.3 (13.6) | 51.8 (12.3) | 51 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 86 | 173
  Male | 91 | 92 | 183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 12
  Not Hispanic or Latino | 162 | 162 | 324
  Unknown or Not Reported | 13 | 7 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 47 | 56 | 103
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 114 | 106 | 220
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 13 | 24
Number of participants with conditioning regimen intensity [Count of Participants; unit: Participants] — Conditioning regimen intensity categorized by myeloablative conditioning (MAC) vs RIC/NMA were reported. MAC regimen consisted: Total body irradiation (TBI) ≥ 5 gray (Gy) single dose or ≥ 8 Gy fractionated/oral Busulfan > 8 milligrams per kilogram (mg/kg)/6.4 mg/kg intravenous (IV) (total dose)/treosulfan >30000 milligrams per square meter (mg/m^2)/elphalan >150 mg/m^2/thiotepa ≥10 mg/kg. RIC/NMA: Any regimen that did not meet MAC regimen: Interactive Response Technology (IRT) analysis was used.
  Participants
    MAC | 103 | 103 | 206
    RIC/NMA | 75 | 75 | 150
Number of Participants With Time from first day of hematopoietic cell infusion to randomization [Count of Participants; unit: Participants] — Number of participants with time from first day of hematopoietic cell infusion to randomization categorized as 30 to 60 days vs 61 to 90 days were reported.
  Participants
    30-60 days | 95 | 97 | 192
    61-90 days | 83 | 81 | 164
Presence of MRD [Count of Participants; unit: Participants] — Number of participants with presence versus absence of, or unknown, MRD-4 from the most recent pre-registration BM aspirate was reported. IRT analysis was used. The presence of MRD was considered "Detectable" if log10-transformed overall FLT3/ITD mutation ratio was greater than -4; otherwise, the presence of MRD was considered "Not Detectable.
  Participants
    Present | 34 | 33 | 67
    Absent/Unknown | 144 | 145 | 289

OUTCOME MEASURES:

1. Primary Outcome: Relapse-free Survival (RFS)
Description: RFS was defined as the time from the date of randomization until the date of documented morphological relapse, or death from any cause, whichever occurred first. Morphological relapse was defined as documentation of any of the following events:
  * BM blasts ≥ 5% (not attributable to regenerating BM)
  * Any circulating blasts (not attributable to regenerating BM or growth factors)
  * Presence of extramedullary blast foci per Revised International Working Group (RIWG) criteria
  * The earliest date of any of the relapse event was used for RFS.
Time Frame: From the date of randomization up to 64 months and 22 days
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gilteritinib | Placebo
Number analyzed (Participants) | 178 | 178
months | NA [NA to NA] — Data was not estimable because less than 50% of participants had event (data was estimated using Kaplan-Meier [KM] and it requires at least 50% of event to be able to calculate time using KM). | NA [NA to NA] — Data was not estimable because less than 50% of participants had event (data was estimated using KM and it requires at least 50% of event to be able to calculate time using KM).
Statistical Analysis 1: Comparison: Gilteritinib vs Placebo; Stratification factors were conditioning regimen intensity MAC vs RIC/NMA, time from transplant to randomization (30 to 60 days vs 61 to 90 days), and the presence of MRD (present vs absent/unknown) based on the pre-transplant BM aspirate; Test type: Superiority; p = 0.0518, Log Rank; Hazard Ratio (HR) = 0.679, 95% CI 2-sided [0.459 to 1.005]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization until the date of death from any cause (death date - first dose date + 1). For a Participant who were not known to have died by the end of study follow-up, OS was censored at the date of last contact (date of last contact - first dose date + 1).
Time Frame: From the date of randomization up to 64 months and 22 day
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gilteritinib | Placebo
Number analyzed (Participants) | 178 | 178
months | NA [NA to NA] — Data was not estimable because less than 50% of participants had event (data was estimated using KM and it requires at least 50% of event to be able to calculate time using KM). | NA [NA to NA] — Data was not estimable because less than 50% of participants had event (data was estimated using KM and it requires at least 50% of event to be able to calculate time using KM).
Statistical Analysis 1: Comparison: Gilteritinib vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4394, Log Rank; Hazard Ratio (HR) = 0.846, 95% CI 2-sided [0.554 to 1.293]

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE)
Description: An Adverse event (AE) was any untoward medical occurrence in a participant administered a study drug, and which did not have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of a medicinal product, whether considered related to the medicinal product.
  TEAE defined as an AE event observed through 30 days after the last dose.
Time Frame: From the date of randomization through 30 days after the last dose, up to 25 months and 22 days
Population: Safety Analysis Population: consisted of all participants who took at least 1 dose of study drug (gilteritinib or placebo).
Measure: Number; unit: participants
Arm/Group | Gilteritinib | Placebo
Number analyzed (Participants) | 178 | 177
participants | 175 | 162

4. Secondary Outcome: Karnofsky Performance Status Scores
Description: KPS scores of participants were reported. KPS was a standard way of measuring ability of cancer participants to perform ordinary tasks. It was 11 level score which ranged between 0-100%. 100 =Normal, no complaints, no evidence of disease 90 =Able to carry on normal activity, minor signs or symptoms of disease 80 =Normal activity with effort, some signs or symptoms of disease 70 =Care for self, unable to carry on normal activity or to do work 60 =Required occasional assistance but was able to care for most of his needs 50 =Required considerable assistance & frequent medical care 40 =Disabled, required special care & assistance 30 = Severely disabled, hospitalization indicated, although death not imminent 20 =Very sick, hospitalization necessary, active supportive treatment necessary 10 =moribund fatal processes progressing rapidly 0 =Dead.
Time Frame: Baseline, month 24
Population: Safety Analysis Population with available data was analyzed.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Gilteritinib | Placebo
Number analyzed (Participants) | 174 | 169
unit on a scale
  Baseline | 84.20 (10.65) | 84.73 (10.69)
  Month 24: number analyzed (Participants) | 93 | 96
  Month 24 | 93.12 (8.34) | 91.67 (9.48)

5. Secondary Outcome: Percentage of Participants With Non-relapse Mortality (NRM)
Description: NRM was defined as death from any cause other than relapse or disease progression (DP). Relapse was defined as documentation of any of the following events:
  * BM blasts ≥ 5% (not attributable to regenerating BM)
  * Any circulating blasts (not attributable to regenerating BM or growth factors)
  * Presence of extramedullary blast foci per RIWG criteria
  * The earliest date of any of the relapse event were used for RFS. DP: >=20% increase in sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline, sum must also be absolute increase of >=5 mm. Unequivocal progression of existing non-target lesions. Appearance of at least 1 new lesion. Incidence of NRM was estimated using the cumulative incidence function, treating relapse/progression as a competing risk.
Time Frame: From the date of randomization up to 64 months and 22 days
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib | Placebo
Number analyzed (Participants) | 178 | 178
percentage of participants | 13.6 [8.9 to 19.2] | 6.6 [3.5 to 11.0]
Statistical Analysis 1: Comparison: Gilteritinib vs Placebo; Based on Fine & Gray's model adjusting for conditioning regimen intensity (MAC vs RIC/NMA), time from transplant to randomization (30-60 days vs 61-90 days) & presence of MRD (present vs absent/indeterminate) based on the pre-transplant BM aspirate; Test type: Superiority; p = 0.0209, Fine-Grays Model; Hazard Ratio (HR) = 2.3080, 95% CI 2-sided [1.1352 to 4.6922]

6. Secondary Outcome: Event-free Survival (EFS)
Description: EFS: Time from date of randomization until documented relapse, or premature discontinuation of treatment or initiation of other anti-leukemic treatment or death from any cause, whichever occurred first.
  Relapse was defined as documentation of any of following events:
  * BM blasts ≥ 5% (not attributable to regenerating BM)
  * Any circulating blasts (not attributable to regenerating BM or growth factors)
  * Presence of extramedullary blast foci per RIWG criteria
  * The earliest date of any of relapse event were used for RFS.
  Anti-leukemic treatment was defined as hypomethylating agents, chemotherapy, oral anticancer agents, Donor lymphocyte infusion (DLI) or cellular therapies given because of detectable disease, not meeting R-IWG criteria for relapse.
Time Frame: From the date of randomization up to 64 months and 22 days
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gilteritinib | Placebo
Number analyzed (Participants) | 178 | 178
months | NA [19.65 to NA] — Data was not estimable because less than 50% of participants had event (data was estimated using KM and it requires at least 50% of event to be able to calculate time using KM). | NA [15.05 to NA] — Data was not estimable because less than 50% of participants had event (data was estimated using KM and it requires at least 50% of event to be able to calculate time using KM).
Statistical Analysis 1: Comparison: Gilteritinib vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.6417, Log Rank; Hazard Ratio (HR) = 0.930, 95% CI 2-sided [0.686 to 1.261]

7. Secondary Outcome: Percentage of Participants With Treatment Emergent Acute Graft vs. Host Disease (aGVHD)
Description: The cumulative incidence at 6 months after randomization of grades II-IV and grades III-IV aGVHD were reported, treating death prior to aGVHD as the competing risk. It was graded according to diagnosis and severity scoring used by the Blood and Marrow Transplant Clinical Trials Network (BMT CTN). The acute GVHD algorithm calculated the grade based on the organ (skin, gastrointestinal (GI)and liver) stage and etiology/biopsy reported on the weekly GVHD form. Grade I aGVHD was defined as Skin stage of 1-2 and stage 0 for both GI and liver organs. Grade II aGVHD was stage 3 of skin, or stage 1 of GI, or stage 1 of liver. Grade III is stage 2-4 for GI, or stage 2-3 of liver. Grade IV was stage 4 of skin, or stage 4 of liver. Grade IV was the worst outcome. Treatment emergent was defined as an event observed through 30 days after the last dose.
Time Frame: From the date of randomization up to 6 months
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib | Placebo
Number analyzed (Participants) | 178 | 178
percentage of participants
  aGVHD II to IV | 16.5 [11.3 to 22.5] | 19.2 [13.6 to 25.6]
  aGVHD III to IV | 5.9 [3.0 to 10.1] | 4.1 [1.8 to 7.9]
Statistical Analysis 1: Comparison: Gilteritinib vs Placebo; aGVHD II to IV: Based on Fine and Gray's model adjusting for conditioning regimen intensity (MAC vs RIC/NMA), time from transplant to randomization (30-60 days vs 61-90 days) & presence of MRD (present vs absent/indeterminate) based on the pre-transplant BM aspirate; Test type: Superiority; p = 0.6410, Fine-Grays model; Hazard Ratio (HR) = 0.8938, 95% CI 2-sided [0.5574 to 1.4330]
Statistical Analysis 2: Comparison: Gilteritinib vs Placebo; aGVHD III to IV: Based on Fine and Gray's model adjusting for conditioning regimen intensity (MAC vs RIC/NMA), time from transplant to randomization (30-60 days vs 61-90 days) & presence of MRD (present vs absent/indeterminate) based on the pre-transplant BM aspirate; Test type: Superiority; p = 0.4128, Fine-Grays model; Hazard Ratio (HR) = 1.4254, 95% CI 2-sided [0.6103 to 3.3289]

8. Secondary Outcome: Percentage of Participants With Treatment Emergent Chronic GVHD at 12 Months
Description: Chronic GVHD was graded according to diagnosis and severity scoring from the National Institute of Health (NIH) 2014 Consensus Criteria. Eight organs - skin, mouth, liver, upper and lower gastrointestinal, esophagus, lung, eye, and joint/fascia were scored on a 0-3 scale to reflect degree of chronic GVHD involvement, where 0 = no involvement/no symptoms & 3 indicated the worst symptom. This system staged severity in each individual organ, and then a global score defined as mild, moderate or severe, based on number of organs involved and organ severity score was calculated. The cumulative incidence of chronic GVHD (mild, moderate, severe) at 12 months after randomization was reported, treating death prior to chronic GVHD as the competing risk. Treatment emergent was defined as an event observed through 30 days after the last dose.
Time Frame: From the date of randomization up to 12 months
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib | Placebo
Number analyzed (Participants) | 178 | 178
percentage of participants | 57.0 [48.5 to 64.6] | 48.1 [39.5 to 56.2]
Statistical Analysis 1: Comparison: Gilteritinib vs Placebo; Based on Fine and Gray's model adjusting for conditioning regimen intensity (MAC vs RIC/NMA), time from transplant to randomization (30-60 days vs 61-90 days) & presence of MRD (present vs absent/indeterminate) based on the pre-transplant BM aspirate; Test type: Superiority; p = 0.1725, Fine-Grays Model; Hazard Ratio (HR) = 1.2360, 95% CI 2-sided [0.9116 to 1.6757]

9. Secondary Outcome: Percentage of Participants With Treatment Emergent Chronic GVHD at 24 Months
Description: Chronic GVHD was graded according to diagnosis and severity scoring from the NIH 2014 Consensus Criteria. Eight organs- skin, mouth, liver, upper and lower gastrointestinal, esophagus, lung, eye, and joint/fascia are scored on a 0-3 scale to reflect degree of chronic GVHD involvement where 0 = no involvement/no symptoms & 3 indicated the worst symptom. This system staged severity in each individual organ, and then a global score defined as mild, moderate or severe, based on number of organs involved and organ severity score was calculated. The cumulative incidence of chronic GVHD (mild, moderate, severe) at 24 months after randomization was reported, treating death prior to chronic GVHD as the competing risk. Treatment emergent was defined as an event observed through 30 days after the last dose.
Time Frame: From the date of randomization up to 24 months
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib | Placebo
Number analyzed (Participants) | 178 | 178
percentage of participants | 61.9 [53.3 to 69.4] | 51.8 [42.9 to 59.9]
Statistical Analysis 1: Comparison: Gilteritinib vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.1725, Fine-Grays Model; Hazard Ratio (HR) = 1.2360, 95% CI 2-sided [0.9116 to 1.6757]

10. Secondary Outcome: Percentage of Participants With FMS-like Tyrosine Kinase 3/Internal Tandem Duplication (FLT3/ITD) Minimal Residual Disease (MRD)
Description: The presence of MRD was considered Detectable in participants who were FLT3/ITD MRD undetectable prior to randomization if log10-transformed overall FLT3/ITD mutation ratio greater than -4 otherwise presence of MRD was considered Not Detectable. Participants who had detectable FLT3/ITD MRD prior to randomization were considered eradicated if log10-transformed overall FLT3/ITD mutation ratio ≤ -4. Incidence of MRD Eradication and Detection were estimated using the cumulative incidence function, treating death during MRD assessment period without documentation of MRD event as competing risk.
Time Frame: From the date of randomization up to 64 months and 22 days
Population: ITT population with available data was analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib | Placebo
Number analyzed (Participants) | 165 | 162
percentage of participants
  MRD Eradication: number analyzed (Participants) | 8 | 10
  MRD Eradication | 80 [4.7 to 98.4] | NA [NA to NA] — Data was not estimable because no participants in Placebo group were followed up to 1 year (cumulative incidence function requires at least 1 participant to calculate the cumulative incidence rate).
  MRD 10^-4 Detection | 7.1 [3.4 to 12.4] | 9.2 [5.0 to 15.0]
Statistical Analysis 1: Comparison: Gilteritinib vs Placebo; MRD Eradication; Test type: Superiority; p = 0.2029, Fine-Grays Model; Hazard Ratio (HR) = 3.4537, 95% CI 2-sided [0.5126 to 23.2687]
Statistical Analysis 2: Comparison: Gilteritinib vs Placebo; MRD 10^-4 Detection; Test type: Superiority; p = 0.4077, Fine-Grays Model; Hazard Ratio (HR) = 0.7073, 95% CI 2-sided [0.3116 to 1.6055]

11. Secondary Outcome: Percentage of Participants With Relapse
Description: Cumulative incidence of relapse was reported, treating death in remission as a competing risk. Relapse was defined as documentation of any of the following events:
  * BM blasts ≥ 5% (not attributable to regenerating BM)
  * Any circulating blasts (not attributable to regenerating BM or growth factors)
  * Presence of extramedullary blast foci per RIWG criteria
  * The earliest date of any of the relapse event were used for RFS.
Time Frame: From the date of randomization up to 64 months and 22 days
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib | Placebo
Number analyzed (Participants) | 178 | 178
percentage of participants | 12.4 [7.9 to 17.8] | 26.7 [20.3 to 33.5]
Statistical Analysis 1: Comparison: Gilteritinib vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.001, Fine-Grays Model; Hazard Ratio (HR) = 0.3729, 95% CI 2-sided [0.2243 to 0.6199]

12. Secondary Outcome: Percentage of Participants With Treatment Emergent Infection by Severity.
Description: Severity of Infection was assessed based on the following criteria:
  Grade 1-Mild Asymptomatic or mild symptoms, clinical or diagnostic observations noted intervention not indicated.
  Grade 2-Moderate Local or noninvasive intervention indicated. Grade 3-Severe Medically significant but not immediately life threatening, hospitalization or prolonged hospitalization. Grade 4-Life Threatening Life threatening consequences, urgent intervention indicated.
  Grade 5-Death related to the AE. Cumulative incidence of grade 3 to 5 infections were reported, treating death (grade 5) as a competing event. Treatment emergent was defined as an event observed through 30 days after the last dose.
Time Frame: From the date of randomization through 30 days after the last dose, up to 25 months and 22 days
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gilteritinib | Placebo
Number analyzed (Participants) | 178 | 178
percentage of participants | 39.6 [31.3 to 47.8] | 27.2 [19.9 to 35.0]
Statistical Analysis 1: Comparison: Gilteritinib vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0568, Fine-Grays model; Hazard Ratio (HR) = 1.4848, 95% CI 2-sided [0.9886 to 2.2300]

ADVERSE EVENTS:
Time Frame: All-cause mortality: From the date of randomization up to 64 months and 22 days Adverse events: From the date of randomization through 30 days after the last dose, up to 25 months and 22 days
Description: Safety Analysis Population. All-cause mortality and serious and other adverse events was reported for all randomized participants who received actual dose of study drug during the study. Therefore, 1 participant randomized to placebo actually received gilteritinib, hence, was included under gilteritinib arm. One participant randomized to gilteritinib arm did not receive any treatment. Serious and other adverse events was reported up to 30 days after last dose.
Arm/Group | Gilteritinib | Placebo
All-Cause Mortality (participants affected / at risk) | 42/178 | 44/177
Serious Adverse Events (participants affected / at risk) | 92/178 | 81/177
Other Adverse Events (participants affected / at risk) | 175/178 | 169/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilteritinib (N=178) | Placebo (N=177)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (6) | 2 (3)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 0 (0)
Antithrombin III deficiency (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Polyserositis (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (5) | 4 (4)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute graft versus host disease (Immune system disorders) | 19 (24) | 22 (27)
Acute graft versus host disease in liver (Immune system disorders) | 0 (0) | 1 (1)
Chronic graft versus host disease (Immune system disorders) | 10 (10) | 8 (8)
Graft versus host disease (Immune system disorders) | 1 (1) | 0 (0)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 (0) | 1 (1)
Graft versus host disease in liver (Immune system disorders) | 0 (0) | 1 (1)
Graft versus host disease in lung (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1 (1) | 0 (0)
Central nervous system infection (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0)
Cystitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 16 (20) | 6 (7)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 3 (5) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 3 (4) | 0 (0)
Viral haemorrhagic cystitis (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (5) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Large granular lymphocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leukaemic retinopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Motor neurone disease (Nervous system disorders) | 1 (1) | 0 (0)
Myelitis transverse (Nervous system disorders) | 1 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Somatic symptom disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 6 (8) | 4 (4)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Vulvovaginal adhesion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Miscarriage of partner (Social circumstances) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Adenoviral upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Clostridial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus enterocolitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter sepsis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Epstein-Barr viraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 3 (3) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 2 (2) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Genital infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 2 (2) | 2 (2)
Oesophageal infection (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 2 (4) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 6 (6) | 3 (3)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection fungal (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viraemia (Infections and infestations) | 1 (1) | 0 (0)
Viral sepsis (Infections and infestations) | 3 (3) | 0 (0)
Viral skin infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilteritinib (N=178) | Placebo (N=177)
Anaemia (Blood and lymphatic system disorders) | 30 (36) | 20 (24)
Neutropenia (Blood and lymphatic system disorders) | 23 (30) | 11 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 22 (29) | 13 (14)
Dry eye (Eye disorders) | 19 (21) | 21 (21)
Abdominal pain (Gastrointestinal disorders) | 11 (13) | 11 (13)
Constipation (Gastrointestinal disorders) | 20 (22) | 12 (14)
Diarrhoea (Gastrointestinal disorders) | 44 (55) | 30 (48)
Dry mouth (Gastrointestinal disorders) | 22 (26) | 15 (17)
Nausea (Gastrointestinal disorders) | 38 (48) | 40 (47)
Vomiting (Gastrointestinal disorders) | 24 (34) | 28 (34)
Fatigue (General disorders) | 30 (40) | 28 (29)
Non-cardiac chest pain (General disorders) | 10 (11) | 1 (1)
Oedema peripheral (General disorders) | 28 (30) | 22 (27)
Pyrexia (General disorders) | 16 (20) | 16 (20)
Alanine aminotransferase increased (Investigations) | 33 (44) | 22 (26)
Aspartate aminotransferase increased (Investigations) | 29 (40) | 21 (24)
Blood alkaline phosphatase increased (Investigations) | 15 (18) | 13 (13)
Blood creatine phosphokinase increased (Investigations) | 33 (41) | 3 (3)
Blood creatinine increased (Investigations) | 17 (22) | 12 (21)
Blood lactate dehydrogenase increased (Investigations) | 9 (11) | 0 (0)
Neutrophil count decreased (Investigations) | 49 (64) | 17 (43)
Platelet count decreased (Investigations) | 32 (44) | 17 (21)
White blood cell count decreased (Investigations) | 22 (31) | 8 (8)
Decreased appetite (Metabolism and nutrition disorders) | 11 (12) | 18 (26)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (15) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 9 (10) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 17 (23) | 4 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 13 (17) | 12 (25)
Hypophosphataemia (Metabolism and nutrition disorders) | 9 (14) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (15) | 12 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (19) | 8 (9)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 (13) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 18 (19) | 9 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (17) | 6 (6)
Dizziness (Nervous system disorders) | 24 (34) | 14 (15)
Headache (Nervous system disorders) | 19 (23) | 13 (17)
Neuropathy peripheral (Nervous system disorders) | 9 (10) | 4 (5)
Paraesthesia (Nervous system disorders) | 9 (10) | 7 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (9) | 2 (2)
Anxiety (Psychiatric disorders) | 10 (10) | 4 (4)
Insomnia (Psychiatric disorders) | 14 (15) | 17 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 33 (40) | 30 (39)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 13 (15)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 9 (11)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (13)
Dry skin (Skin and subcutaneous tissue disorders) | 14 (16) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (13) | 13 (15)
Rash (Skin and subcutaneous tissue disorders) | 10 (13) | 16 (22)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 (13) | 9 (11)
Hypertension (Vascular disorders) | 28 (35) | 13 (21)
Acute graft versus host disease (Immune system disorders) | 67 (90) | 64 (91)
Chronic graft versus host disease (Immune system disorders) | 94 (156) | 77 (131)
Cytomegalovirus viraemia (Infections and infestations) | 8 (10) | 12 (16)
Influenza (Infections and infestations) | 11 (11) | 5 (5)
Pneumonia (Infections and infestations) | 8 (9) | 10 (12)
Upper respiratory tract infection (Infections and infestations) | 21 (25) | 22 (34)
Viral upper respiratory tract infection (Infections and infestations) | 18 (21) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT02997202/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT02997202/SAP_001.pdf